CLINICAL TRIAL: NCT01644955
Title: Intracerebral Convection Enhanced Delivery of Carboplatin for Treatment of Recurrent High-grade Gliomas
Brief Title: Carboplatin in Treating Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Elder (Other)
Responsible Party: Sponsor-Investigator, James Elder, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10151; NCI-2012-01057 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Recurrent Adult Brain Tumor
Keywords: Gliomas; Carboplatin
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Brain Neoplasms; Glioma | interventions — Carboplatin; Surgical Procedures, Operative; Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carboplatin) (Experimental): Patients will undergo surgery, which includes tumor resection and catheter placement, in the operating room and then receive carboplatin administered intracerebrally by convection enhanced delivery.
  Interventions: Drug: carboplatin; Procedure: Surgery

INTERVENTIONS:
Drug: carboplatin — Carboplatin in a volume of 54 ml will be administered intracerebrally by convection enhanced delivery
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Procedure: Surgery — Patients will undergo surgery, which includes tumor resection and catheter placement, in the operating room.
  Other Names: craniotomy

SUMMARY:
This study is being done to evaluate the toxicity and safety of carboplatin administered by convection enhanced delivery into the tumor in patients with high grade glial neoplasms. This study is a dose escalating study, (the dose of the study drug is increased at set time points). Carboplatin is in a class of drugs known as platinum-containing compounds; it slows or stops the growth of cancer cells in your body. Convection enhanced delivery involves placing one or more catheters into the brain and delivering chemotherapy through those catheters directly into the brain

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the maximum tolerated dose and define the toxicity profile of carboplatin delivered intracerebrally via convection enhanced delivery (CED) for patients with high grade glial neoplasms.

SECONDARY OBJECTIVES:

I. Examine the efficacy as defined by six-month progression free survival (PFS), median progression free survival, overall survival, and the radiographic response rate.

II. Evaluate the drug distribution.

OUTLINE: This is a phase I, dose-escalation study.

Patients undergo craniotomy and then receive carboplatin intracerebrally via convection-enhanced delivery (CED) over 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have progressive disease for which craniotomy and tumor resection is recommended as treatment
* Patients must sign a consent form indicating that they are aware of the investigational nature of the study; the informed consent form will indicate that the patient has been made aware of all other appropriate therapies
* Patients with histologically confirmed grade III or IV astrocytoma, oligoastrocytoma, and oligodendroglioma who are at first or second recurrence
* Patients require an initial diagnosis of a malignant glioma as outlined in the inclusion criteria which must be confirmed at the treating facility
* Patients must have unequivocal evidence of tumor progression by magnetic resonance imaging (MRI) performed no longer than 28 days prior to study registration
* Patients must have pathologically confirmed recurrence at the time of catheter placement
* Patients must be on a stable or decreasing dexamethasone dosage for at least 1 week prior to baseline MRI
* Patients must have been treated previously with radiation therapy and treatment must have been completed at least 8 weeks prior to surgery for catheter implantation
* Last dose of cytotoxic chemotherapy must have been at least 4 weeks (6 weeks for nitrosoureas) prior to catheter placement; patients are eligible if they received bevacizumab or other anti-vascular endothelial growth factor (VEGF) therapies, although the most recent dose must be at least 6 weeks prior to catheter placement
* Patients previously treated with stereotactic radiosurgery, stereotactic radiotherapy, brachytherapy, Gliadel wafers or other intratumoral chemotherapy are eligible
* Patients must have recovered from all prior therapy
* Patients must have a life expectancy of >= 3 months and a Karnofsky performance status >= 60 Leukocytes >= 3,000/mcL Absolute neutrophil count >= 1,500/mcL Platelets >= 100,000/mcL Hemoglobin >= 9 g/dL Serum calcium =< 12.0 mg/dL Total serum bilirubin < institutional upper limit of normal (ULN) Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN Creatinine < 1.5 X institutional ULN
* Women of child bearing years must have a negative pregnancy test (serum or urine) within 1 week of study entry; men and women of reproductive potential must agree to use an effective contraceptive method including one of the following: surgical sterilization (tubal ligation for women or vasectomy for men); approved hormonal contraceptives (such as birth control pills, Depo-Provera or Lupron Depro); barrier methods (such as condom or diaphragm) used with a spermicide cream or an intrauterine device (IUD)
* Patient or designated individuals with durable medical power of attorney must give written informed consent prior to any study-specific procedures being implemented
* Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients with infratentorial, multifocal, or pathologically confirmed cerebrospinal fluid (CSF) disseminated tumor
* Patients that have been treated with > 3 prior chemotherapy regimens
* Pregnant or lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Patients who have a history of bleeding disorders including congenital or acquired coagulopathies
* Known acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition or other acquired or congenital disorder of the immune system
* Patients with unstable or serious concurrent illness including, but not limited to, ongoing or active infections requiring IV antibiotics or psychiatric illness/social situations that would limit compliance with study requirements are ineligible; (if patient has a stable chronic infection requiring oral antibiotics, the patient may be treated at the investigators discretion; however a clinical note must include the justification regarding the safety of treating the patient)
* Patients who have received any other investigational agent in a 28-day period prior to enrollment in this study
* Patients whose tumors are located less than 2 cm from the ventricles
* Patients taking greater than 12 mg daily of dexamethasone
* Prior invasive malignancy that is not low-grade glioma, glioblastoma or gliosarcoma (except non-melanomatous skin cancer or carcinoma in situ of the cervix) unless the patient has been disease free and off therapy for that disease for a minimum of 3 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Establish maximum tolerated dose and define toxicity profile | 72 hours after maximal medical therapy is initiated
  The toxicity profile of carboplatin delivered intracerebrally via convection enhanced delivery (CED) for patients with high grade glial neoplasms. The maximum tolerated dose (MTD) of infused carboplatin may then be incorporated into future clinical studies.

SECONDARY OUTCOMES:
Six month progression free survival defined as the proportion of patients with stable disease at 6 months from surgery | Time between surgery and earliest sign of disease progression or death, assessed up to 6 months
Median progression free survival | Time between surgery and earliest sign of disease progression or death, assessed up to 2 years
Radiographic response rate | Up to 2 years
Overall survival | Time from surgery until death, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Elder, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu